CLINICAL TRIAL: NCT05540990
Title: The Effectiveness of Robot Assisted Gait Training In Children With Cerebral Palsy: Randomized Comparative Trial
Brief Title: Robot Assisted Gait Training In Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Birkan Sonel Tur, Clinical Professor, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: İ5-310-21
Record Dates: First submitted 2022-09-02; First posted 2022-09-15 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Cerebral Palsy; Physical Therapy; Robotic Rehabilitation; Motor Skills Disorders
Keywords: Cerebral Palsy, Robot assisted gait training, Gait
MeSH Terms: conditions — Cerebral Palsy; Motor Skills Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic assisted gait training (RAGT) + conventional physiotherapy (CPt) group (Experimental): This group will receive 15 sessions of robot-assisted gait training (two or three times per week with a maximum of 45 minutes each) and conventional physiotherapy, which is individually customized to the needs of the child and usually consists of 2-3 sessions of physiotherapy per week.
  Interventions: Device: Robot assisted gait training; Other: Conventional physiotherapy
- Conventional physiotherapy (CPt) group (Active Comparator): This group will receive conventional physiotherapy, which is individually customized to the needs of the child and usually consists of 2-3 sessions of physiotherapy per week.
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Device: Robot assisted gait training — 15 sessions of robot-assisted gait training (two times per week with a maximum of 45 minute each).
  Arms: Robotic assisted gait training (RAGT) + conventional physiotherapy (CPt) group
Other: Conventional physiotherapy — individually customized to the needs of the child and usually consists of 2-3 sessions of physiotherapy per week.

SUMMARY:
Cerebral Palsy (CP) is considered a neurological disorder caused by a non-progressive brain injury or malformation that occurs while the child's brain is under development. CP primarily affects body movement and muscle coordination. Robot assisted gait training (RAGT) is considered to be a promising approach for improving gait related gross motor function of children and youth with CP.

There is weak and inconsistent evidence regarding the use of RAGT for children with gait disorders. Further research is required with increased numbers and with relevant outcome measures to both confirm the effectiveness and clarify training schedules.

The aim of this research project is to investigate the effectiveness of robot assisted gait training on improvements of functional gait parameters in children with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is a disorder of posture and movement due to a defect in the immature brain. There is evidence that locomotor therapy for regaining walking capacity using the principle of enhancing neuroplasticity by task-specific training is effective in the rehabilitation process of patients with central gait disorders. The use of a robotic device assists in achieving and maintaining physiological walking pattern for extended periods of therapy. The use of robotic devices as an alternative treatment to improve the gait function in patients with CP has increased.

This is a prospective, randomized comparative trial (RCT). This study is designed to compare the effectiveness of conventional physical therapy (CPt) and robot assisted gait training (RAGT) on gait related motor skills of children with cerebral palsy.

Children aged 5 to 18 years with GMFCS Level 2-4, bilateral or unilateral spastic CP are accepted into this study. Participants are randomly assigned to receive CPt or RAGT + CPt.

All two intervention groups will receive 2-3 sessions of CPt per week over 6-8 weeks. CPt sessions are individually customized to the needs of the child.

The participants of RAGT + CPt group also receive 15 sessions of RAGT (2-3 times per week with a maximum of 45 minute each).

ELIGIBILITY:
Inclusion Criteria:

* GMFCS Level 2-4
* Bilateral or unilateral spastic CP
* Able to follow instructions and communicate pain or discomfort
* Have a passive range of motion (ROM) of hips and knees within minimum range requirement for robotic assisted training (hip and knee flexion contracture ≤10°, and knee valgus ≤40°)
* Not having participated in another robotic assisted training regime within the previous 6 months
* Able to participate in a minimum of 30 minutes robotic assisted training session
* Able to commit to attendance of two to three times weekly for 15 sessions (to support the primary efficacy analysis)

Exclusion Criteria:

* Botulinum toxin type A injection within 3 months
* Orthopedic surgery on the lower extremity (muscle surgery within the last 9 months, bone surgery within 12 months)
* Bone fractures, open skin lesions, or circulatory problems
* Vision and hearing impairments that affect participation in robotic assisted training
* Epilepsy resistant to medication
* Cardiopulmonary instability
* Use of a baclofen pump

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Change in GMFM-88 D Item | baseline, 8 weeks, 14 weeks and 20 weeks
  The Gross Motor Function Measure (GMFM) is an assessment tool designed and evaluated to measure changes in gross motor function over time or with intervention in children with cerebral palsy. GMFM-88 is a measure developed to evaluate the gross motor function changes in CP children. It has five components: lying and rolling, sitting, kneeling and crawling, standing, and walking. D dimension is for Standing abilities. The score of each dimension is expressed as a percentage of the maximum score.
  There is a scoring system with each item scored as 0, 1, 2, 3, or "not tested". A scoring key of 0 - does not initiate, 1 - initiates, 2 - partially completes, and 3 - completed, is used.
  It takes between 20-25 minutes to be completed.
Change in GMFM-88 E Item | baseline, 8 weeks, 14 weeks and 20 weeks
  The Gross Motor Function Measure (GMFM) is an assessment tool designed and evaluated to measure changes in gross motor function over time or with intervention in children with cerebral palsy. GMFM-88 is a measure developed to evaluate the gross motor function changes in CP children. It has five components: lying and rolling, sitting, kneeling and crawling, standing, and walking. E dimension is for Walking, Running & Jumping abilities. The score of each dimension is expressed as a percentage of the maximum score.
  There is a scoring system with each item scored as 0, 1, 2, 3, or "not tested". A scoring key of 0 - does not initiate, 1 - initiates, 2 - partially completes, and 3 - completed, is used.
  It takes between 20-25 minutes to be completed.

SECONDARY OUTCOMES:
Change in 6 Minute Walk Test | baseline, 8 weeks, 14 weeks and 20 weeks
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Change in 10 Meter Walk Test | baseline, 8 weeks, 14 weeks and 20 weeks
  The 10 Metre Walk Test is a performance measure used to assess walking speed in meters per second over a short distance.
Change in Modified Ashworth Scale | baseline, 8 weeks, 14 weeks and 20 weeks
  The modified Ashworth scale is the most universally accepted clinical tool used to measure the increase of muscle tone.
Change in Goal Attainment Scale (GAS) | baseline, 8 weeks, 14 weeks and 20 weeks
  The GAS methodology is congruent with the client-centered occupational therapy philosophy because GAS provides a means to identify intervention outcomes that are specifically relevant to individuals and their families.
Change in Pediatric Quality of Life Inventory (PedsQL) 3.0 Cerebral Palsy Module (Parent Form) | baseline, 8 weeks, 14 weeks and 20 weeks
  The PedsQL 3.0 CP module is questionnaire designed to assess the quality of life in children with cerebral palsy. The 35-item PedsQL 3.0 CP Module encompasses seven scales: (1) Daily Activities (9 items); (2) School Activities (4items); (3) Movement and Balance (5 items); (4) Pain andHurt (4 items); (5) Fatigue (4 items); (6) Eating Activities (5items); and (7) Speech and Communication (4 items). A 5-point response scale is utilized across child self-report for ages 8 to 18 years and parent proxy-report (0=never a problem; 1=almost never a problem;2=sometimes a problem; 3=often a problem; 4=almostalways a problem).

CONTACTS AND LOCATIONS:
Overall Officials: Birkan Sonel Tur, Prof, Principal Investigator — Ankara University
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)